CLINICAL TRIAL: NCT02796469
Title: Statistical Analysis Plan for an Individual Patient Data Meta-analysis of Ten Clinical Trials Comparing Drug Therapy in Patients With Severe Alcoholic Hepatitis
Brief Title: Meta-Analysis of Drug Therapy in Patients With Severe Alcoholic Hepatitis
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: MA_2016-01
Record Dates: First submitted 2016-05-31; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Alcoholic Hepatitis; Alcoholic Liver Disease
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Diseases, Alcoholic | interventions — Pentoxifylline; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pentoxifylline + Corticosteroid: Association of treatment by pentoxifylline and corticosterone during 28 days
  Interventions: Drug: Pentoxifylline; Drug: Corticosteroid
- Corticosteroid: treatment by corticosteroid during 28 days
  Interventions: Drug: Corticosteroid; Drug: Placebo
- Pentoxifylline: treatment by pentoxifylline during 28 days
  Interventions: Drug: Pentoxifylline; Drug: Placebo
- Placebo

INTERVENTIONS:
Drug: Pentoxifylline
  Groups: Pentoxifylline; Pentoxifylline + Corticosteroid
Drug: Corticosteroid
  Groups: Corticosteroid; Pentoxifylline + Corticosteroid
Drug: Placebo
  Groups: Corticosteroid; Pentoxifylline

SUMMARY:
In the specific setting of the evaluation of corticosteroids, pentoxifylline of their combination in severe alcoholic hepatitis, only meta-analysis combining individual data is able to provide detailed information from each individual with severe alcoholic hepatitis assessed by a DF ≥ 32. The need for such an approach is confirmed by the fact that in both univariate and multivariate analyses, truth survival is lower for conclusions from meta-analysis of the literature than for conclusions derived from non-meta-analyses.

The present study is a meta-analysis of individual data from RCTs restricted to patients with a DF ≥ 32. The primary endpoint will be to compare 28-day survival of patients receiving either corticosteroids, or pentoxifylline or their combination to those of patients not receiving them adjusted on the independent prognostic factors at baseline.

The secondary endpoints will be: a) assessment of response to the assigned treatment using the Lille model; b) analysis of 6-month survival according to allocated therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients included in 10 randomized controlled trials testing either corticosteroids alone, or pentoxifylline alone or their combination have been published.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe alcoholic hepatitis assessed by Discriminant Function (DF) ≥32.
Sampling Method: Non-Probability Sample
Enrollment: 1974 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | at 28 days, after the first administration of treatment

SECONDARY OUTCOMES:
Lille Model Score | at day 7, after the first administration of treatment
  Lille model evaluate to therapy and will be analyzed as dichotomous outcome (<0.45 vs. ≥0.45), ordinal outcome (≤0.16 vs. 0.16-0.56 vs. ≥ 0.56) and continuous outcome (after log-transformation) and will be restricted to patients with a dosage of bilirubin at day 7 after initiation of assignment treatment.
Biological measure : Bilirubin | at day 7, at day 28
  evaluate of bilirubin during treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Mathurin, MD, PhD, Principal Investigator — University Hospital, Lille

IPD SHARING:
Plan to Share IPD: Undecided